CLINICAL TRIAL: NCT01380301
Title: Treatment of Bolivian Cutaneous Leishmaniasis With a Combination of Short Courses of Miltefosine and Antimony
Brief Title: Treatment of Cutaneous Leishmaniasis With a Combination of Miltefosine and Antimony
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low efficacy rates
Sponsor: Foundation Fader (Other)
Collaborators: AB Foundation (Other)
Responsible Party: JAIME SOTO, Foundation Fader
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-Bol-01
Record Dates: First submitted 2009-01-28; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Leishmaniasis; Miltefosine; Antimony; Therapy
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — miltefosine; Antimony

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Miltefosine and Antimony (Experimental): Miltefosine 1,5 to 2,5 mg x k x d during 14 days simultaneously with meglumine antimoniate 20 mg x kg x d during 10 days
  Interventions: Drug: Miltefosine and antimony
- Miltefosine alone (Active Comparator): Miltefosine 1,5 to 2,5 mg x kg x d during 14 days
  Interventions: Drug: Miltefosine alone

INTERVENTIONS:
Drug: Miltefosine and antimony — Short course (half of each drug) administered simultaneously
  Arms: Miltefosine and Antimony
Drug: Miltefosine alone — short course (half)
  Arms: Miltefosine alone

SUMMARY:
Cutaneous leishmaniasis is endemic in the New World and, until recently, the standard treatment was pentavalent antimony. The cure rate for L panamensis in Colombia is 91%-93% and the cure rate in Bolivia is also 90%. Nevertheless, pentavalent antimonials have the disadvantages of multiple injections and mild-moderate clinical toxicity all of which are particularly unpleasant for a moderate clinical problem such as cutaneous leishmaniasis.

The oral agent Miltefosine has now been shown to be as effective as antimony in Colombia and Bolivia (91 and 92% respectively). Side effects seen in patients with cutaneous disease that can be specifically attributed to the drug are nausea and vomiting of mild grade in approximately 25% of patients, and low-grade elevation of creatinine also in approximately 25% of patients. A further disadvantage of miltefosine is that regimens shorter than 4 weeks have not been evaluated for cutaneous disease.

Combination therapy is now being used for many infectious diseases, such as tuberculosis, malaria, and HIV. Combination therapy offers the potential of preventing drug resistance, because organisms resistant to one of the drugs may be susceptible to the other drug; and also the potential to diminish drug therapy duration and thus side effects. These two potential benefits to some extent contradict each other: preventing resistance is best done if full courses of both drugs is used; diminishing therapy duration means using less than the full course of each drug. The optimum combination regimen is one in which sufficient amounts of both drugs are used to have high efficacy, yet the amounts are as low as possible to spare patients unnecessarily long courses of drug.

In the present protocol, the combination of a half-course of miltefosine and a half-course of antimony will be evaluated for efficacy and tolerance. The combination of miltefosine and antimony is chosen because these are now the two standard agents in Bolivia, and in vitro the combination was additive to mildly synergistic against a standard leishmania strain.

ELIGIBILITY:
Inclusion Criteria:

* Parasitological confirmation
* at least 1 lesion must be ulcerative
* No specific antileishmanial therapy during the previous six months

Exclusion Criteria:

* Concomitant diseases such as Tuberculosis, HIV, diabetes, renal failure, liver disease
* abnormalities CTC 2 in blood, liver, kidney test or EKG

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Healing of ulcers | 45 days

SECONDARY OUTCOMES:
Clinical findings and Laboratory parameters in normal ranges | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: JONATHAN BERMAN, MD, PhD, Study Director — AB Foundation
Locations (1):
- Hospital Local, La Paz, La Paz Department, Bolivia